CLINICAL TRIAL: NCT02056015
Title: A Phase 1, First-in-Human, Single-Dose, Open-Label, Positron Emission Tomography (PET) Imaging Study of [68Ga]MLN6907 in Patients With Metastatic Colorectal Carcinoma.
Brief Title: A Phase I Study of MLN6907 in Patients With Metastatic Colorectal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C35001
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Imaging of Solid Gastrointestinal Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [68Ga]MLN6907 (Experimental)
  Interventions: Drug: [68Ga]MLN6907

INTERVENTIONS:
Drug: [68Ga]MLN6907 — IV Administration of [68Ga]MLN6907 on Day 1

SUMMARY:
This study is a first-in-human (FIH), single-dose, open-label, phase 1 study designed to assess the safety, pharmacokinetics (PK), distribution, and radiation dosimetry of [68Ga]MLN6907 after a single intravenous (IV) administration. Patients with Metastatic Colorectal Carcinoma who are scheduled for resection of liver metastases as part of their treatment plan will be eligible for enrollment.

ELIGIBILITY:
Inclusion Criteria

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Male or female patients 18 years or older.
* Must be diagnosed with colorectal cancer (CRC) with liver metastasis and eligible and scheduled for resection of liver metastases as part of their standard of care treatment plan. The planned surgery must occur greater than 14 days after the day of imaging.
* Patients must consent to provide the sponsor with tumor tissue samples from their resected liver metastases.
* Easter Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Female patients who are post menopausal, surgically sterile, or agree to practice effective methods of contraception from the time of signing the informed consent form through 60 days after the dose of [68Ga]MLN6907 or agree to practice true abstinence.
* Male patients who agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the dose of [68Ga]MLN6907 or agree to practice true abstinence.
* Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
* Suitable venous access for the study-required, blood sampling (ie, including PK sampling)
* Adequate hepatic function as defined in the protocol.
* Adequate renal function as defined in the protocol.
* Hemoglobin ≥ 9 g/dL.
* Recovery from all adverse effects from prior antitumor therapy to at least Common Terminology Criteria for Adverse Events (CTCAE) (V4.03) Grade 1.

Exclusion Criteria

Patients meeting any of the following exclusion criteria are not to be enrolled in the study.

* Female patients who are lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before the first dose of [68Ga]MLN6907.
* Any serious medical or psychiatric illness, condition, or personal circumstance, including severe claustrophobia, severe dyspnea, severe back pain, etc., that, in the judgment of the investigator or project clinician, might potentially interfere with the procedures required in this study.
* Involvement in an investigative radioactive or other research procedure within 4 weeks prior to administration of [68Ga]MLN6907.
* Major surgery within 14 days prior to administration of [68Ga]MLN6907 5. Serious infection (viral, bacterial, or fungal) within 14 days before administration of [68Ga]MLN6907 or evidence of active infection during screening.
* Life-threatening illness unrelated to cancer.
* Clinically significant central nervous system (CNS) metastases.
* Known inflammatory bowel disease.
* Known hepatitis B surface antigen-positive or known or suspected active hepatitis C infection (testing not required).
* History of any hypersensitivity to any component of [68Ga]MLN6907.
* Symptomatic cardiac disease, including ventricular dysfunction, coronary artery disease, or arrhythmias, if this would, in the opinion of the investigator or project clinician, interfere with assessment of efficacy or safety of [68Ga]MLN6907.
* Admission or evidence of addictive disorders (eg, illicit drug use, drug abuse, or alcohol abuse) that would limit compliance with study requirements.
* Inability to lie flat for the duration of image acquisition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs), serious AEs (SAEs), assessments of clinical laboratory values, and vital sign measurements | Duration of study up to 26 months
Human organ and whole body absorbed dose values from organ kinetic quantification of [68Ga]MLN6907 uptake and clearance | Day 1

SECONDARY OUTCOMES:
Expert visual rating of [68Ga]MLN6907 liver tumor uptake and quantitative measurement of tumor-to-background (normal liver, muscle, etc.) ratio for each liver tumor | Duration of study up to 26 months
Time-activity curves for each liver tumor region of interest (ROI) and kinetic curves of the ratio of each liver tumor to background (including for normal liver, muscle, and blood); determination of the time for the maximum ratio for each tumor lesion | Duration of study up to 26 months
Plasma [68Ga]MLN6907 and MLN6907 drug substance precursor PK parameters and quantification of GCC levels in liver metastases | Day 1
  PK parameters include single-dose maximum (peak) concentration (Cmax), single-dose time to reach maximum (peak) concentration (Tmax), terminal disposition half-life (t1/2), and area under the plasma concentration versus time curve (AUC).
Correlate tumor uptake of [68Ga]MLN6907 measured by PET and the level of guanylyl cyclase C (GCC) expression in tumor lesions from surgical specimens , for tumors in individual patients and for aggregated liver tumors across patients | Duration of study up to 26 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (2):
- Iowa City, Iowa, United States
- Alburquerque, New Mexico, Mexico